CLINICAL TRIAL: NCT00474760
Title: Phase 1, Open Label, Multiple Dose Escalation Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of CP 751,871 In Patients With Advanced Solid Tumors
Brief Title: Study Of Anti-IGF-IR CP-751,871 In Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4021010
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-10

CONDITIONS: Sarcoma, Ewing's
MeSH Terms: conditions — Sarcoma, Ewing | interventions — figitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: CP-751,871

INTERVENTIONS:
Drug: CP-751,871 — Currently dosing at 20 mg/kg, IV on day 1 of each 28 day cycle until progression or unacceptable toxicity

SUMMARY:
This is a phase 1 study of anti-IGF-IR CP-751,871 in patients with solid tumors currently enrolling patients 9 years old and older with Ewing's sarcoma family of tumors (Ewing's, PNET and Askin's).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ewing's sarcoma family tumors

Exclusion Criteria:

* Concurrent treatment with any other anti tumor agents

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-08; Primary Completion 2011-01 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (2):
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
- Pfizer Investigational Site, Sutton, Surrey, United Kingdom

REFERENCES:
- [Derived] Asmane I, Watkin E, Alberti L, Duc A, Marec-Berard P, Ray-Coquard I, Cassier P, Decouvelaere AV, Ranchere D, Kurtz JE, Bergerat JP, Blay JY. Insulin-like growth factor type 1 receptor (IGF-1R) exclusive nuclear staining: a predictive biomarker for IGF-1R monoclonal antibody (Ab) therapy in sarcomas. Eur J Cancer. 2012 Nov;48(16):3027-35. doi: 10.1016/j.ejca.2012.05.009. Epub 2012 Jun 7. PMID 22682017
- [Derived] Olmos D, Postel-Vinay S, Molife LR, Okuno SH, Schuetze SM, Paccagnella ML, Batzel GN, Yin D, Pritchard-Jones K, Judson I, Worden FP, Gualberto A, Scurr M, de Bono JS, Haluska P. Safety, pharmacokinetics, and preliminary activity of the anti-IGF-1R antibody figitumumab (CP-751,871) in patients with sarcoma and Ewing's sarcoma: a phase 1 expansion cohort study. Lancet Oncol. 2010 Feb;11(2):129-35. doi: 10.1016/S1470-2045(09)70354-7. Epub 2009 Dec 23. PMID 20036194

RESULTS

PARTICIPANT FLOW:
Groups:
- Figitumumab 3 mg/kg: Figitumumab 3 milligram/kilogram (mg/kg) was supplied as a liquid solution administered as an intravenous (IV) infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for dose escalation cohort.
- Figitumumab 6 mg/kg: Figitumumab 6 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for dose escalation cohort.
- Figitumumab 10 mg/kg: Figitumumab 10 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for dose escalation cohort.
- Figitumumab 20 mg/kg: Figitumumab 20 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for dose escalation cohort.
- Figitumumab 20 mg/kg RP2D: Figitumumab 20 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for recommended Phase 2 dose [RP2D] extension cohort.
- Figitumumab 20 mg/kg RP2D ACC+Sarcoma: Figitumumab 20 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for RP2D adrenocortical carcinoma [ACC] and sarcoma extension cohort.
- Figitumumab 20 mg/kg RP2D ESFT: Figitumumab 20 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (4 weeks in duration) for RP2D Ewing's sarcoma family of tumors [ESFT] extension cohort.
Period: Overall Study
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D | Figitumumab 20 mg/kg RP2D ACC+Sarcoma | Figitumumab 20 mg/kg RP2D ESFT
Started | 3 | 3 | 3 | 3 | 13 | 29 | 11
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not Completed | 3 | 3 | 3 | 3 | 12 | 29 | 10
Not completed — Death | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 7 | 0
Not completed — Laboratory abnormality | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Other | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive disease | 3 | 2 | 3 | 2 | 8 | 20 | 7
Not completed — Terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Figitumumab 3 mg/kg: Figitumumab 3 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for dose escalation cohort.
- Figitumumab 20 mg/kg RP2D: Figitumumab 20 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for RP2D extension cohort.
- Figitumumab 20 mg/kg RP2D ACC+Sarcoma: Figitumumab 20 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for RP2D ACC and sarcoma extension cohort.
- Figitumumab 20 mg/kg RP2D ESFT: Figitumumab 20 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (4 weeks in duration) for RP2D ESFT extension cohort.
- Total: Total of all reporting groups
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D | Figitumumab 20 mg/kg RP2D ACC+Sarcoma | Figitumumab 20 mg/kg RP2D ESFT | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 13 | 29 | 11 | 65
Age, Customized [Number; unit: participants]
  Less than (<) 70 years | 3 | 3 | 3 | 3 | 13 | 28 | 11 | 64
  Equal to or greater than (>=) 70 years | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 0 | 1 | 13 | 3 | 21
  Male | 2 | 1 | 2 | 3 | 12 | 16 | 8 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 150 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 150 days after the last administration of study drug
Population: All enrolled participants who started treatment.
Measure: Number; unit: participants
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D | Figitumumab 20 mg/kg RP2D ACC+Sarcoma | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 13 | 29 | 11
participants
  AEs | 3 | 3 | 3 | 3 | 13 | 29 | 11
  SAEs | 2 | 1 | 3 | 1 | 5 | 17 | 5

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) in Cycle 1
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: All participants treated who had at least 1 of the pharmacokinetic (PK) parameters of primary interest. N=number of participants evaluable for the outcome measure. Summaries for figitumumab 20 mg/kg RP2D, and figitumumab 20 mg/kg RP2D ACC and sarcoma extension cohorts were combined into 1 reporting group: figitumumab 20 mg/kg RP2D every 3 weeks.
Measure: Mean (Standard Deviation); unit: milligram/liter (mg/L)
Groups:
- Figitumumab 20 mg/kg RP2D Every 3 Weeks: Figitumumab 20 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for RP2D, and RP2D ACC and sarcoma extension cohorts.
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 34 | 9
milligram/liter (mg/L) | 57.77 (2.658) | 134.7 (31.754) | 211.0 (59.808) | 463.0 (97.964) | 457.5 (135.68) | 392.0 (90.308)

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) in Cycle 4
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: All participants treated who had at least 1 of the PK parameters of primary interest in extension cohorts. N=number of participants evaluable for the outcome measure. Summaries for figitumumab 20 mg/kg RP2D, and figitumumab 20 mg/kg RP2D ACC and sarcoma extension cohorts were combined into 1 reporting group: figitumumab 20 mg/kg RP2D every 3 weeks.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 16 | 6
mg/L | 697.2 (165.40) | 650.8 (169.92)

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) in Cycle 1
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: All participants treated who had at least 1 of the PK parameters of primary interest. N=number of participants evaluable for the outcome measure. Summaries for figitumumab 20 mg/kg RP2D, and figitumumab 20 mg/kg RP2D ACC and sarcoma extension cohorts were combined into 1 reporting group: figitumumab 20 mg/kg RP2D every 3 weeks.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 34 | 9
hours | 8.361 (13.552) | 1.147 (0.117) | 1.043 (0.075) | 0.678 (0.558) | 9.394 (28.527) | 3.441 (7.718)

5. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) in Cycle 4
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 16 | 6
hours | 7.541 (16.343) | 4.840 (9.436)

6. Secondary Outcome: Plasma Decay Half-Life (t1/2) in Cycle 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 2 | 1 | 3 | 1 | 8 | 2
hours | 203.0 (7.071) | 226.0 | 252.3 (56.713) | 227.0 | 259.6 (80.500) | 319.0 (8.485)

7. Secondary Outcome: Plasma Decay Half-Life (t1/2) in Cycle 4
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 5 | 3
hours | 386.0 (172.16) | 479.7 (163.59)

8. Secondary Outcome: Time to Reach Last Quantifiable Concentration (Tlast) in Cycle 1
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 34 | 9
hours | 501.0 (4.583) | 443.0 (96.995) | 523.7 (41.041) | 498.3 (1.155) | 509.5 (100.13) | 666.7 (3.082)

9. Secondary Outcome: Time to Reach Last Quantifiable Concentration (Tlast) in Cycle 4
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 16 | 6
hours | 418.7 (227.37) | 743.7 (100.81)

10. Secondary Outcome: Systemic Clearance (CL) in Cycle 1
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliliter/day/kilogram (mL/day/kg)
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 2 | 1 | 3 | 1 | 7 | 2
milliliter/day/kilogram (mL/day/kg) | 6.435 (2.199) | 3.600 | 4.807 (2.059) | 4.990 | 3.846 (1.101) | 3.155 (0.559)

11. Secondary Outcome: Systemic Clearance (CL) in Cycle 4
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 9 | 6
mL/day/kg | 2.576 (0.484) | 2.612 (1.112)

12. Secondary Outcome: Concentration at End of Infusion (Cendinf) in Cycle 1
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 33 | 9
mg/L | 57.50 (3.081) | 134.7 (31.754) | 211.0 (59.808) | 463.0 (97.964) | 434.3 (94.278) | 386.3 (96.496)

13. Secondary Outcome: Concentration at End of Infusion (Cendinf) in Cycle 4
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 16 | 6
mg/L | 685.0 (167.15) | 650.3 (170.80)

14. Secondary Outcome: Volume of Distribution (Vz) in Cycle 1
Description: Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliliter/kilogram (mL/kg)
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 2 | 1 | 3 | 1 | 7 | 2
milliliter/kilogram (mL/kg) | 78.00 (24.183) | 49.00 | 70.47 (25.733) | 68.10 | 59.34 (14.360) | 60.35 (9.122)

15. Secondary Outcome: Volume of Distribution (Vz) in Cycle 4
Description: as for outcome 14
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 5 | 3
mL/kg | 61.98 (20.741) | 89.17 (47.461)

16. Secondary Outcome: Volume of Distribution at Steady State (Vss) in Cycle 1
Description: Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the Vz at steady-state.
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 2 | 1 | 3 | 1 | 7 | 2
mL/kg | 75.05 (20.011) | 47.90 | 68.80 (23.477) | 66.90 | 59.27 (14.765) | 61.65 (6.435)

17. Secondary Outcome: Volume of Distribution at Steady State (Vss) in Cycle 4
Description: as for outcome 16
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 5 | 3
mL/kg | 60.84 (19.694) | 86.07 (42.133)

18. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) in Cycle 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligram*hour/liter (mg*hr/L)
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 31 | 9
milligram*hour/liter (mg*hr/L) | 10900 (3005.0) | 27500 (5656.9) | 43900 (19630) | 89430 (11904) | 107900 (36398) | 102700 (25300)

19. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) in Cycle 4
Description: Area under the plasma concentration time-curve from zero to the last measured concentration
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 16 | 6
mg*hr/L | 166500 (77400) | 214500 (67592)

20. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] in Cycle 1
Description: Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0 - ∞).
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 2 | 1 | 3 | 1 | 7 | 2
mg*hr/L | 11910 (4094.1) | 40000 | 57770 (28167) | 96300 | 136000 (47622) | 154500 (27577)

21. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to 504 Hours (21 Days) (AUC504) in Cycle 1
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: All participants treated who had at least 1 of the PK parameters of primary interest in all cohorts except ESFT extension cohort. N=number of participants evaluable for the outcome measure. Summaries for figitumumab 20 mg/kg RP2D, and RP2D ACC and sarcoma extension cohorts were combined into 1 reporting group: 20 mg/kg RP2D every 3 weeks.
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D Every 3 Weeks
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 31
mg*hr/L | 10900 (3005.0) | 27500 (5656.9) | 43170 (20124) | 89430 (11904) | 104000 (32547)

22. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to 504 Hours (21 Days) (AUC504) in Cycle 4
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Figitumumab 20 mg/kg RP2D Every 3 Weeks
Number analyzed (Participants) | 9
mg*hr/L | 193100 (40001)

23. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to 672 Hours (28 Days) (AUC672) in Cycle 1
Time Frame: Cycle 1: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: All participants treated who had at least 1 of the PK parameters of primary interest in RP2D ESFT extension cohort. N=number of participants evaluable for the outcome measure
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 9
mg*hr/L | 102400 (25227)

24. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to 672 Hours (28 Days) (AUC672) in Cycle 4
Time Frame: Cycle 4: 0 (predose), 1, 24 and 72 hours, 7 and 14 days postdose
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Figitumumab 20 mg/kg RP2D ESFT
Number analyzed (Participants) | 6
mg*hr/L | 207200 (72334)

25. Secondary Outcome: Human Anti-human Antibodies (HAHA) Levels
Description: HAHA were indicators of immunogenicity to figitumumab.
Time Frame: 30 minutes predose in Cycles 1 up to 61, and last scheduled follow-up visit (up to 150 days from the last dose of study drug)
Population: Per protocol, the presence of HAHA would only be evaluated for those samples with plasma figitumumab concentrations below the limit of quantification (BLQ). Since none of the postdose samples in the study had figitumumab concentrations BLQ, therefore no sample was analyzed for HAHA.
Groups:
- Figitumumab 3, 6, 10, 20 mg/kg: Figitumumab 3, 6, 10, or 20 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration for dose escalation, RP2D extension, and RP2D ACC and sarcoma extension cohorts, 4 weeks in duration for RP2D ESFT extension cohort).
Arm/Group | Figitumumab 3, 6, 10, 20 mg/kg
Number analyzed (Participants) | 0

26. Secondary Outcome: Number of Circulating Tumor Cells (CTCs)
Description: Quantification of CTCs using an automated microscope system
Time Frame: 30 minutes predose in all cycles (up to 17); 1, 3, 7, and 14 days postdose in Cycle 1 for dose escalation and RP2D extension cohorts; and also 1 day postdose in Cycle 4 for RP2D extension cohort
Population: Pretreatment CTCs were detected in an insufficient number of participants to analyze for any treatment effect on this pharmacodynamic biomarker.
Groups:
- Figitumumab 3, 6, 10, 20 mg/kg: Figitumumab 3, 6, 10, or 20 mg/kg was supplied as a liquid solution administered as an IV infusion over 2.5 hours (plus or minus 15 minutes) on Day 1 of each cycle (3 weeks in duration) for dose escalation and RP2D extension cohorts.
Arm/Group | Figitumumab 3, 6, 10, 20 mg/kg
Number analyzed (Participants) | 0

27. Secondary Outcome: Number of Insulin-like Growth Factor 1 Receptor (IGF-1R) Positive CTCs
Description: Quantification of IGF-IR positive CTCs using an automated microscope system
Time Frame: as for outcome 26
Population: Pretreatment IGF-1R positive CTCs were detected in an insufficient number of participants to analyze for any treatment effect on this pharmacodynamic biomarker.
Arm/Group | Figitumumab 3, 6, 10, 20 mg/kg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Figitumumab 3 mg/kg | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg | Figitumumab 20 mg/kg RP2D | Figitumumab 20 mg/kg RP2D ACC+Sarcoma | Figitumumab 20 mg/kg RP2D ESFT
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 3/3 | 1/3 | 5/13 | 17/29 | 5/11
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 13/13 | 29/29 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 3 mg/kg (N=3) | Figitumumab 6 mg/kg (N=3) | Figitumumab 10 mg/kg (N=3) | Figitumumab 20 mg/kg (N=3) | Figitumumab 20 mg/kg RP2D (N=13) | Figitumumab 20 mg/kg RP2D ACC+Sarcoma (N=29) | Figitumumab 20 mg/kg RP2D ESFT (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Disease progression (General disorders) | 1 | 1 | 3 | 1 | 2 | 8 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood culture positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 3 mg/kg (N=3) | Figitumumab 6 mg/kg (N=3) | Figitumumab 10 mg/kg (N=3) | Figitumumab 20 mg/kg (N=3) | Figitumumab 20 mg/kg RP2D (N=13) | Figitumumab 20 mg/kg RP2D ACC+Sarcoma (N=29) | Figitumumab 20 mg/kg RP2D ESFT (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2 | 3 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delayed puberty (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Miosis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 9 | 4
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 6 | 5 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 8 | 13 | 4
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 3 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 6 | 6 | 7
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Crepitations (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 3 | 6 | 12 | 7
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Activated partial thromboplastin time abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 5 | 6 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 0 | 7 | 7 | 1
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 4 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 4 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood magnesium increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Blood uric acid increased (Investigations) | 1 | 1 | 1 | 1 | 3 | 5 | 1
Body temperature (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 2 | 0 | 5 | 7 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 2 | 3 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Pulse abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 2 | 2 | 5 | 14 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3 | 5 | 8 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 6 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 7 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 5 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 6 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 4 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 7 | 4
Hyporeflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phantom pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 3 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3 | 4 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0
Alopecia totalis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1

LIMITATIONS AND CAVEATS:
The study was completed and 2 participants in figitumumab 20 mg/kg RP2D ESFT group were transitioned to compassionate figitumumab treatment as investigators judged they were receiving benefit from the protocol therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.